CLINICAL TRIAL: NCT00289601
Title: Research Evaluation to Study Individuals Who Show Thromboxane Or P2Y12 Receptor Resistance
Brief Title: Randomized Study of Aspirin Resistant Patients Undergoing Angioplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor support withdrawn
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RESISTOR
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Angioplasty
Keywords: aspirin; clopidogrel; resistance; angioplasty; percutaneous coronary intervention; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: eptifibatide

SUMMARY:
This study is a randomized, double-blind, multi-center study designed to compare differences in rates of myonecrosis (measured as an elevation of CK-MB ratio ≥ 2 times ULN) within 24 hours following low-medium risk percutaneous coronary intervention (PCI) in aspirin or clopidogrel non-responsive patients who are randomized to heparin with or without eptifibatide therapy during PCI. The primary objective of this study is to determine if the use of eptifibatide is associated with a significant difference in post-PCI myonecrosis (measured as an elevation of CK-MB ratio ≥ 2 times upper limit of normal [ULN]) within 24 hours of low-medium risk PCI in patients who are aspirin or non-responsive as determined by VerifyNow Aspirin and P2Y12 testing.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if the use of eptifibatide is associated with a significant difference in post-PCI myonecrosis (measured as an elevation of CK-MB ratio ≥ 2 times upper limit of normal [ULN]) within 24 hours of low-medium risk PCI in patients who are aspirin or clopidogrel non-responsive as determined by VerifyNow Aspirin and P2Y12 testing.

Secondary study objectives will include an assessment of safety. These safety determinations will be determined by monitoring the rates of MACE (defined as death, MI, ischemic [non-hemorrhagic] stroke and urgent revascularization by repeat PCI or CABG), bleeding events, rate of bailout procedures performed, elevations of CK-MB ratio (in the range of 3 to 5 times ULN and greater than 5 times ULN) and elevations of troponin I.

This study is a randomized, double-blind, multi-center study designed to compare differences in rates of myonecrosis (measured as an elevation of CK-MB ratio ≥ 2 times ULN) within 24 hours following low-medium risk percutaneous coronary intervention (PCI) in aspirin or clopidogrel non-responsive patients who are randomized to heparin with or without eptifibatide therapy during PCI. All subjects must also be pretreated with clopidogrel (300-600 mg) at least 2 hours before PCI. Study subjects will be randomized to either eptifibatide and unfractionated heparin or unfractionated heparin and placebo. Study subject randomization in aspirin non-responsive patients will be stratified based upon clopidogrel responsiveness.

ELIGIBILITY:
Inclusion Criteria:

Patients with coronary artery disease will be eligible for the study. Inclusion criteria are:

Patient is 21 years or older. Patient is scheduled to undergo low-medium risk percutaneous coronary intervention in native coronary vessels.

Patient self-reports that he/she has received aspirin ≥ 81 mg at least 4 hours prior to study screening.

Patient is defined as aspirin non-responsive based upon results of the VerifyNow™ Aspirin test, defined as an aspirin reaction units (ARU) > 475.

Patient is defined as clopidogrel non-responsive based upon the results of the VerifyNow P2Y12 test, defined as less than 20% inhibition.

Patient will be treated with 300- 600 mg of clopidogrel at least two hours before the intervention.

All patients will provide written informed consent, and the study protocol will be approved by the IRB of the participating centers.

Patient is male, or is a non-pregnant female.

Exclusion Criteria:

Patient has a known allergic reaction to the study medication. Patient has been diagnosed with a myocardial infarction within the prior 7 days.

Patient has unstable angina, defined as dynamic, ischemic ECG changes (ST-segment elevation, ST-segment depression, or T-wave inversion) at rest.

Patient has rest pain with left bundle branch block. Note: In a patient with rest pain and abnormal ECG that is believed to be non-acute (i.e., STTW abnormalities secondary to LVH, digoxin, or prior remote infarction), a second electrocardiogram 30 min apart is required to establish that these changes are non-dynamic and not indicative of active ischemia.

The target lesion(s) is located in a venous bypass graft. The patient has a chronic occlusion (present for longer than 3 months). The target lesion(s) has visible thrombus (by angiography). The patient has had a suspected aortic dissection. Patient has left ventricular ejection (LVEF) < 30%. Patient was receiving oral anticoagulation therapy.

Patient received any of the following drugs during 7 days prior to enrollment:

* any GP IIb/IIIa inhibitor
* ticlopidine
* dipyridamole
* cilostazol (Pletal) Patient has received non-steroidal anti-inflammatory drugs (NSAIDS), or any steroidal drugs 24 hours prior to enrollment.

Patient has been diagnosed with any stroke within the prior 3 months. Patient has active bleeding or bleeding diathesis. Patient has experienced trauma or major surgery in the preceding month. Patient has severe, uncontrolled hypertension (systolic blood pressure of more than 180 mm Hg).

Patient's creatinine > 2.0 mg/dl prior to PCI. Patient has a hemoglobin level of less than 10.0 g per deciliter or a hematocrit below 30 percent.

Patient has a platelet count of less than 100,000 per cubic millimeter or more than 600,000 per cubic millimeter.

Of note, patients on chronic clopidogrel will only be eligible for VerifyNow P2Y12 testing. Clopidogrel non-responsiveness in this group will be defined as < 20% inhibition

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2006-03; Study Completion 2007-12

PRIMARY OUTCOMES:
The primary endpoint is the incidence of myonecrosis, defined as an elevation in creatinine kinase - myocardial band (CK-MB) > 2 x IU/ml above the institution's upper limit of normal within 24 hours following low-medium risk PCI.

SECONDARY OUTCOMES:
Incidence of CK-MB elevation >3x ULN
Incidence of CK-MB elevation to 3-5x ULN
Incidence of CK-MB elevation >5x ULN
Incidence of troponin I > 0.1ng/ml
MACE rates reported at discharge, 30 days and 6 months. (MACE is defined as a composite endpoint of death, MI, ischemic (non-hemorrhagic) stroke, and urgent target vessel revascularization)
Rate of bail-out use of eptifibatide/placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Simon, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States